CLINICAL TRIAL: NCT04102722
Title: A Prospective, Single-Center, Feasibility Study Assessing the Safety and Performance of the Multi-Modal UltraSound Tomography (MUST) Device in Identifying Malignant Breast Lesions as an Adjunct to Mammography
Brief Title: Safety and Performance of the Multi-Modal UltraSound Tomography (MUST) Device in Breast Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Transonic Imaging, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MUST-02-001
Record Dates: First submitted 2019-06-11; First posted 2019-09-25 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer Screening
Keywords: tomography; ultrasound; mammogram; breast

STUDY DESIGN:
Intervention Model Description: All enrolled subjects will receive breast cancer screening with mammography and MUST
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Experimental): All enrolled subjects will undergo breast cancer screening with mammography and the MUST device
  Interventions: Device: MUST device

INTERVENTIONS:
Device: MUST device — Imaging with MUST device

SUMMARY:
This is a single-center, pilot study being conducted to evaluate the safety and performance of the investigational device (MUST) in detecting malignant lesions in breast tissue.

DETAILED DESCRIPTION:
This is a single-center, prospective, pilot study in which all enrolled subjects will receive the same screening mammography procedures (i.e., 3D mammography plus MUST).

Subjects will have between 1 and 4 clinic visits. The number of visits will be based upon the mammography and MUST findings, and whether additional procedures, such as MRI, biopsy, or a repeat MUST are warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Female subject scheduled for routine screening mammogram
2. Not currently pregnant or breastfeeding
3. Age 40 to 74 years, inclusive
4. Weight less than 115 kg
5. Able to provide written informed consent
6. Willing to comply with study protocol and follow-up recommendations.

Exclusion Criteria:

1. Breast implants
2. Signs or symptoms of breast disease including changes in the size or shape of breast tissue, palpable lump, bloody or spontaneous clear nipple discharge, and/or eczema of the nipple
3. Weeping rash, open wounds, or unhealed sores on the breast
4. Bilateral mastectomy or unilateral mastectomy
5. Unable to lay prone on the scan table for up to 16 minutes
6. Unable to have breast positioned into the MUST device
7. Any breast surgeries in the past 12 months
8. History of cancer diagnosis and/or treatment in the past 5 years.
9. Unable or unwilling to undergo MRI if indicated

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1333 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with true positive (malignant) breast lesions confirmed by biopsy | 14 days
  Sensitivity of MUST plus mammography versus mammography alone
Number of subjects with false positive (benign) breast lesions confirmed by biopsy | 14 days
  Specificity of MUST plus mammography versus mammography alone

SECONDARY OUTCOMES:
Number of true positive and false positive breast lesions categorized by BI-RADS breast density category as determined by the screening mammogram | 14 days
  Assess the sensitivity and specificity by BI-RADS breast density category as determined by the Visit 1 mammogram, for MUST plus mammography vs mammography alone
For subjects who undergo biopsy, comparison of MUST results with biopsy results | 60 days
  In the subpopulation of subjects who undergo biopsy, the concordance of MUST with biopsy will be estimated
For subjects test positive on mammography (initial BI-RADS score of 0 followed by an additional imaging BI-RADS score of 4 or 5) who undergo biopsy, comparison of MUST and MRI results with biopsy results | 60 days
  In the subpopulation of subjects who test positive on mammography (BI-RADS score of 4 or 5) and have a biopsy, sensitivity and specificity will be assessed and compared between MUST and MRI and biopsy results
Number of subjects with true positive and false positive breast lesions at the 6 month follow up (if applicable) and the 12 month follow up phone call. | 12 months
  The co-primary endpoint of overall sensitivity and specificity will be reassessed after subjects have had the opportunity to complete the Month 6 MUST re-evaluation visit, if applicable, and again when all subjects have had the opportunity to complete the Month 12 follow-up phone call to identify events of interval cancer for MUST plus mammography as well as MUST alone
Listing of adverse events experienced by subjects | 6 months
  Evaluate the safety of the MUST device by evaluating the adverse event profile

CONTACTS AND LOCATIONS:
Overall Officials: Tejas Mehta, MD, Principal Investigator — Beth Israel Deaconess Hospital
Locations (1):
- Beth Israel Deaconess Medical Center BreastCare Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided